CLINICAL TRIAL: NCT00517894
Title: Phase 3 Study of Dose-Dense Therapy Versus CHOP in Aggressive Non-Hodgkin's Lymphoma
Brief Title: Dose-Dense Therapy in Aggressive Lymphoma
Status: No longer available | Type: Expanded Access
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Other Study IDs: NHL-5
Record Dates: First submitted 2007-08-15; First posted 2007-08-17 (Estimated); Last update posted 2007-08-17 (Estimated); Status verified 2007-08

CONDITIONS: Lymphoma
Keywords: lymphoma; aggressive; chemotherapy; dose-dense
MeSH Terms: conditions — Lymphoma; Aggression

INTERVENTIONS:
Drug: CEOP/IMVP-Dexa chemotherapy — Cyclophosphamide 750 mg/m2 i.v. d 1, epirubicin 70 mg/m2 i.v d 1, vincristine 1.4 mg/m2 i.v. d 1+8, prednisolone 100 mg p.o. d 1-5, ifosfamide 2000 mg/m2 i.v. d 15-17, etoposide 100 mg/m2 i.v. d 15-17, dexamethasone 40 mg p.o. or i.v. d 15-19, methotrexate 800 mg/m2 i.v. d 22. Mesna was given with ifosfamide, calcium-folinate rescue after methotrexate. Filgrastim was given on days 2-7, 9-12, 18-21, 23-28

SUMMARY:
To investigate if a dose-dense chemotherapy with weekly chemotherapy compared to standard treatment every 3 weeks results in better survival in aggressive non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
Patients are randomized to receive dose-dense CEOP/IMVP-Dexa chemotherapy or standard 3-weekly CHOP.

ELIGIBILITY:
Inclusion Criteria:

* 18 and 70 years of age
* Centrally reviewed, histologically proven diffuse large B-cell, anaplastic large-cell, or peripheral T-cell unspecified
* Measurable disease
* All stages

Exclusion Criteria:

* Lymphoblastic or Burkitt histology
* CNS-disease
* HIV-positive
* pregnant or lactating women
* Pretreatment
* Other malignancy
* Concomitant diseases that forbid chemotherapy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- [Derived] Fridrik MA, Hausmaninger H, Lang A, Drach J, Krieger O, Geissler D, Michlmayr G, Ulsperger E, Chott A, Oberaigner W, Greil R. Dose-dense therapy improves survival in aggressive non-Hodgkin's lymphoma. Ann Hematol. 2010 Mar;89(3):273-82. doi: 10.1007/s00277-009-0811-x. Epub 2009 Aug 20. PMID 19693500